CLINICAL TRIAL: NCT01925183
Title: Response-guided Triple-therapy Using Boceprevir in Combination With PEGIFN/RBV in HIV/HCV-coinfected Patients
Brief Title: Individualized Triple-therapy Using Boceprevir in HIV-positive Patients With Hepatitis C
Acronym: HIVCOBOC-RGT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Markus Peck-Radosavljevic (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Markus Peck-Radosavljevic, Vice-chairman of the Division of Gastroenterology and Hepatology, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIVCOBOC-RGT; 2012-005591-33 (EudraCT Number)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C, Chronic; HIV
Keywords: Boceprevir; HIV/HCV-coinfection; HIV/HCV coinfection; HIV/HCV; Response-guided therapy
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 28 weeks of treatment duration (Experimental): All patients will receive 4 weeks of PEGIFN/RBV lead-in. Patients with undetectable HCV-RNA at treatment week 8 will be treated with 24 weeks of BOC/PEGIFN/RBV triple-therapy resulting in a total treatment duration of 28 weeks.
  Interventions: Drug: Pegylated interferon alpha-2a; Drug: Ribavirin; Drug: Boceprevir
- 48 weeks of treatment duration (Experimental): All patients will receive 4 weeks of PEGIFN/RBV lead-in. Patients with detectable HCV-RNA at treatment week 8 will receive 44 weeks of BOC/PEGIFN/RBV triple-therapy and a total treatment duration of 48 weeks
  Interventions: Drug: Pegylated interferon alpha-2a; Drug: Ribavirin; Drug: Boceprevir

INTERVENTIONS:
Drug: Pegylated interferon alpha-2a — 180mcg once weekly; subcutaneous injection
  Other Names: Pegasys®, Roche
Drug: Ribavirin — 600mg two times daily (BID) (e.g. 3x200mg at 6am, 3x200mg at 6pm) in patients ≥75kg body weight; 2x200mg at 6am and 3x200mg at 6pm in patients <75kg; orally
  Other Names: Copegus®, Roche
Drug: Boceprevir — 800mg three times daily (TID) (e.g. 4x200mg at 6am, 4x200mg at 2pm, 4x200mg at 10pm); orally
  Other Names: Victrelis®, MSD

SUMMARY:
Response-guided triple-therapy with boceprevir (BOC) in combination with pegylated interferon (PEGIFN) and ribavirin (RBV) is the current standard of care for HIV-negative patients infected with hepatitis C genotype (HCV-GT) 1. In contrast, in HIV-positive patients, a fixed treatment duration of 48 weeks is used.

The aim of this study is to assess efficacy and safety of response-guided triple-therapy with BOC in combination with PEGIFN and RBV in HIV-positive patients. Thus, treatment duration will be individualized based on HCV-RNA negativity at treatment week 8 (W8). All patients will receive 4 weeks of PEGIFN/RBV lead-in. Patients with undetectable HCV-RNA at W8 will be treated with 24 weeks of BOC/PEGIFN/RBV triple-therapy resulting in a total treatment duration of 28 weeks, while patients with detectable HCV-RNA at W8 will receive 44 weeks of BOC/PEGIFN/RBV triple-therapy and a total treatment duration of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection (anti-HIV1/2 antibody positive).
* Chronic HCV infection (anti-HCV positive, HCV-RNA detectable for >6 months).
* HCV-GT 1 infection.
* Age ≥18 years and ≤65 years.
* No prior treatment with BOC/PEGIFN/RBV.
* CD4+ cell count >200 cells/µL.
* Stable antiretroviral therapy (ART) including tenofovir/emtricitabine (Truvada®, Gilead) and raltegravir (Isentress®, MSD) with HIV-RNA <50 copies/mL.
* Valid result on transient elastography or liver biopsy within 6 months prior to enrollment.
* Female patients of childbearing potential must agree to use an effective contraceptive during treatment and for 4 months after treatment has been concluded.
* Male patients or their female partners must agree to use an effective contraceptive during treatment and for 7 months after treatment has been concluded.

Exclusion Criteria:

* HCV-GT other than HCV-GT 1.
* Cirrhotic patients (as defined by METAVIR F4 in liver biopsy or liver stiffness >12.3 kPa) with decompensated liver disease (Child-Pugh stage B/C).
* Chronic liver diseases other than hepatitis C virus infection (hepatitis B virus infection: HBsAg positivity, nonalcoholic steatohepatitis, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cystic fibrosis).
* Significant cardiac disease (ejection fraction <40% at echocardiography).
* Significant pulmonary disease (COPD stage GOLD III/IV).
* Significant renal disease (serum creatinine >1.5 mg/dL).
* Subjects taking medication(s) that is/are highly dependent on CYP3A4/5 for clearance, and for which elevated plasma concentrations are associated with serious and/or life-threatening events such as but not limited to, orally administered midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine, and ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine).
* Contraindications for boceprevir (Victrelis®, MSD), pegylated interferon alpha-2a (Pegasys®, Roche) or ribavirin (Copegus®, Roche), as listed in section 4.3 of the respective summary of product characteristics (SmPCs).
* Ongoing alcohol abuse (average daily alcohol consumption >50g).
* Ongoing illicit drug abuse.
* Unwillingness to give written informed consent.
* Pregnancy and breastfeeding.
* Women wishing to become pregnant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Peck-Radosavljevic, MD, Principal Investigator — Division of Gastroenterology and Hepatology, Department of Internal Medicine III, Medical University of Vienna
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine III, Medical University of Vienna, Vienna, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- 28 Weeks of Treatment Duration: All patients will receive 4 weeks of pegylated interferon/ribavirin (PEGIFN/RBV) lead-in. Patients with undetectable hepatitis C virus (HCV)-RNA at treatment week 8 will be treated with 24 weeks of boceprevir (BOC)/PEGIFN/RBV triple-therapy resulting in a total treatment duration of 28 weeks.
  Pegylated interferon alpha-2a: 180mcg once weekly; subcutaneous injection
  Ribavirin: 600mg two times daily (BID) (e.g. 3x200mg at 6am, 3x200mg at 6pm) in patients ≥75kg body weight; 2x200mg at 6am and 3x200mg at 6pm in patients <75kg; orally
  Boceprevir: 800mg three times daily (TID) (e.g. 4x200mg at 6am, 4x200mg at 2pm, 4x200mg at 10pm); orally
Period: Overall Study
Arm/Group | 28 Weeks of Treatment Duration | 48 Weeks of Treatment Duration
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 28 Weeks of Treatment Duration | 48 Weeks of Treatment Duration | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Sustained Virologic Response (SVR12)
Description: Defined as HCV-RNA negativity by a sensitive assay
Time Frame: Follow-up week 12 (FU12)
Measure: Count of Participants; unit: Participants
Arm/Group | 28 Weeks of Treatment Duration | 48 Weeks of Treatment Duration
Number analyzed (Participants) | 3 | 3
Participants | 3 | 2

2. Primary Outcome: Proportions of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline (BL) to Follow-up week 12 (FU12)
Measure: Count of Participants; unit: Participants
Arm/Group | 28 Weeks of Treatment Duration | 48 Weeks of Treatment Duration
Number analyzed (Participants) | 3 | 3
Participants
  Adverse events (AEs) | 3 | 3
  Serious adverse events (SAEs) | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline (BL) to Follow-up week 12 (FU12)
Arm/Group | 28 Weeks of Treatment Duration | 48 Weeks of Treatment Duration
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 28 Weeks of Treatment Duration (N=3) | 48 Weeks of Treatment Duration (N=3)
Abscess soft tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 28 Weeks of Treatment Duration (N=3) | 48 Weeks of Treatment Duration (N=3)
Psoriasis (Immune system disorders) | 1 (1) | 0 (0) — Psoriasis flare-up
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes